CLINICAL TRIAL: NCT02918162
Title: A Phase II Study of Chemotherapy and Immune Checkpoint Blockade With Pembrolizumab in the Perioperative and Maintenance Treatment of Locoregional Gastric or GE Junction Adenocarcinoma.
Brief Title: Perioperative Chemo and Pembrolizumab in Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gulam Manji (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Gulam Manji, Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ9871
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer; Adenocarcinoma of the Gastroesophageal Junction
Keywords: pembrolizumab; adenocarcinoma; gastric cancer; Locoregional gastric adenocarcinoma; Locoregional GE junction adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): All study subjects will receive standard of care chemotherapy regimen for 3 cycles prior to and 3 cycles following surgery in combination with Pembrolizumab with an additional cycle of Pembrolizumab (4 total) in the pre-operative period. Additionally subjects will complete 12 months of maintenance Pembrolizumab (14 additional doses to complete 17 post-operative cycles) following completion of post-operative chemotherapy.
  Standard of care combination chemotherapy regimen has a 21-day cycle.
  Interventions: Drug: Pembrolizumab; Drug: Standard of care chemotherapy regimen

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab dosed IV at 200mg every 21 days per cycle.
  Other Names: KEYTRUDA; MK-3475
Drug: Standard of care chemotherapy regimen — Standard regimen containing at least a platinum and Fluorouracil (5-FU) agent (per National Comprehensive Cancer Network guidelines) - such as Doublet or Triplet chemotherapy with capecitabine, oxaliplatin, and epirubicin (optional) (21 day cycle). Epirubicin can be excluded at the discretion of the treating physician.
  Example:
  Oxaliplatin dosed IV at 130 mg/m2 every 21 days per cycle. Capecitabine dosed orally at 625mg/m2 twice a day daily.
  Other Names: Investigator's choice of of standard regimen

SUMMARY:
This is a non-randomized, multi-site, open-label trial of pembrolizumab and chemotherapy in subjects with gastric or gastroesophageal (GE) junction adenocarcinoma. The purpose of this study is to determine and evaluate the efficacy of combination therapy with immune checkpoint blockade and chemotherapy used in the perioperative period in eradicating micrometastatic disease; and to compare paired tissue and serum samples (pre-treatment and post-treatment) from individually treated patients to explore the immune effects of combination therapy and predictors of response.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common cancers worldwide. Surgical resection is the primary treatment for gastric cancer but most patients present with locally advanced disease and recurrence is common after surgery. Many patients (35%) will have early recurrence within 6-9 months of surgery indicating the need for more aggressive upfront therapy in these subjects. In addition, the majority of patients will ultimately have recurrence and 5 year survival rates are 35-40% despite aggressive therapy.

The ability to combine immunotherapy with pembrolizumab gives the potential to increase therapeutic options while continuing standard of care chemotherapy. The particular use of maintenance therapy may delay or eliminate the growth of residual micrometastatic disease and lead to durable disease control. Additionally, this study provides the foundation for substantial correlative work to define tumor and patient characteristics that may predict for response to pembrolizumab in gastric cancer.

The initial primary outcome of Disease Free Survival (DFS) was changed to pathologic complete response rate (pCR) on November 24, 2020, at which time no formal data analysis had been preformed.

ELIGIBILITY:
Inclusion Criteria:

1. Have previously untreated localized gastric or GE junction adenocarcinoma as defined by T2 or greater primary lesion or the presence of any positive nodes- N+(clinical nodes) without evidence of metastatic disease.
2. Plan to proceed to surgery following peri-operative chemotherapy based on standard staging studies per local practice.
3. Be willing and able to provide written informed consent/assent for the trial. The subject may also provide consent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research.
4. Be at least 18 years of age on day of signing informed consent.
5. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1.
6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
7. Demonstrate adequate organ function as defined below, all screening labs should be performed within 14 days of treatment initiation.

   Adequate Organ Function Laboratory Values
   * Absolute neutrophil count (ANC) ≥1,500 /mcL
   * Platelets ≥100,000 / mcL
   * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
   * Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
   * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
   * Albumin >2.5 mg/dL
   * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   * Creatinine clearance should be calculated per institutional standard.
8. Have a 2D Echocardiogram with left ventricular ejection fraction = or > 45% in order to receive Epirubicin. Subjects with inadequate EF or other contraindication can proceed on study without the use of Epirubicin.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential must be willing to use an adequate method of contraception - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Male subjects of childbearing potential must agree to use an adequate method of contraception - Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids (prednisone 10 mf or equivalent) may be approved after consultation.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had any prior chemotherapy, targeted small molecule therapy, or radiation therapy for their current diagnosis.
6. Has a known additional malignancy that is progressing or requires active treatment within 3 years from registration. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Subjects with a history of prior malignancy diagnosed and treated greater than 3 years form registration may be considered with consultation of the primary investigator.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has known history of prior pneumonitis requiring treatment with steroids, or any evidence of active, non-infectious pneumonitis.
10. Has an active infection requiring systemic therapy which is not expected to have resolved by Cycle 1 Day 1 dosing.
11. Has a history or current evidence of any condition (e.g. known deficiency of the enzyme dihydropyrimidine dehydrogenase [DPD]),, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor-investigator staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific subject.
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gulam Manji, MD, PhD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Haesong Park, St Louis, Missouri
  - Weill Cornell Medical College/ NewYork-Presbyterian, New York, New York
  - Columbia University Medical Center, New York, New York
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Manji GA, Lee S, Del Portillo A, May M, Ana SS, Alouani E, Sender N, Negri T, Gautier K, Ge L, Fan W, Xie M, Sethi A, Schrope B, Tan AC, Park H, Oberstein PE, Shah MA, Raufi AG. Chemotherapy and Immune Checkpoint Blockade for Gastric and Gastroesophageal Junction Adenocarcinoma. JAMA Oncol. 2023 Dec 1;9(12):1702-1707. doi: 10.1001/jamaoncol.2023.4423. PMID 37856106
- See also: Cancer Center's clinical trials online search tool — http://www.hiccc.columbia.edu/ct/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 49 participants signed a consent form, 10 of which were screen failures and 3 of which withdrew consent prior to completion of screening.
Groups:
- Pembrolizumab: All study subjects will receive standard of care chemotherapy regimen for 3 cycles prior to and 3 cycles following surgery in combination with Pembrolizumab with an additional cycle of Pembrolizumab (4 total) in the pre-operative period. Additionally subjects will complete 12 months of maintenance Pembrolizumab (14 additional doses to complete 17 post-operative cycles) following completion of post-operative chemotherapy.
  Standard of care combination chemotherapy regimen has a 21-day cycle.
  Pembrolizumab: Pembrolizumab dosed IV at 200mg every 21 days per cycle.
  Standard of care chemotherapy regimen: Standard regimen containing at least a platinum and Fluorouracil (5-FU) agent (per National Comprehensive Cancer Network guidelines) - such as Doublet or Triplet chemotherapy with capecitabine, oxaliplatin, and epirubicin (optional) (21 day cycle). Epirubicin can be excluded at the discretion of the treating physician.
  Example:
  Oxaliplatin dosed IV at 130 mg/m2 every 21 days per cycle. Capecitabine dosed orally at 625mg/m2 twice a day daily.
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 36
Completed | 34
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Omental Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 65 [25 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate
Description: Number of subjects with absence of viable tumor on surgical resection specimen as determined by local pathology review.
Time Frame: Up to 34 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 34
Participants | 7

2. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from Cyle 1 Day 1 treatment administration to death due to any cause. The 24 month overall survival probability was estimated using the Kaplan-Meier method.
Time Frame: Treatment initiation until death or study end, whichever occurs first (up to approximately 5 years)
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 34
Probability | 80.6 [67.6 to 96.1]

3. Secondary Outcome: Disease Free Survival (DFS)
Description: DFS defined as time from Cycle 1 Day 1 treatment administration to the first documented event of disease progression, disease recurrence following surgery (preferably biopsy proven), or death whichever occurs first. The 24 month DFS probability was estimated using the Kaplan-Meier method.
Time Frame: Treatment initiation to progression, recurrence, death or study end, whichever comes first (up to approximately 5 years)
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 34
Probability | 67.8 [53.1 to 86.6]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Number of subjects with initial RECIST 1.1 measurable disease who have complete response (CR) or partial response (PR) at any time (ORR= CR + PR). CR defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 34 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 34
Participants | 14

ADVERSE EVENTS:
Time Frame: Up to 34 months
Description: Systematic assessment of adverse events: Routine review of and for adverse events at each scheduled visit through investigator assessment and laboratory testing. 36 participants enrolled in the study, one participant withdrew consent, therefore 35 were included in adverse events assessment.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 8/35
Serious Adverse Events (participants affected / at risk) | 9/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=35)
Diarrhea (Gastrointestinal disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Sepsis (Infections and infestations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=35)
Diarrhea (Gastrointestinal disorders) | 20
Fatigue (General disorders) | 23
Peripheral sensory neuropathy (Nervous system disorders) | 20
Nausea (Gastrointestinal disorders) | 19
Anorexia (Metabolism and nutrition disorders) | 11
Vomitting (Gastrointestinal disorders) | 11
Neutrophil count decreased (Investigations) | 10
Anemia (Blood and lymphatic system disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Hypothyroidism (Endocrine disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 4
Platelet count decreased (Investigations) | 4
Adrenal insufficiency (Endocrine disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Chills (General disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 3
Dry mouth (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Headache (Nervous system disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 2
Paresthesia (Nervous system disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Weight loss (Investigations) | 3
Allergic reaction (Immune system disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Flu like symptoms (General disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain (General disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 2
White blood cell decreased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Body odor (Skin and subcutaneous tissue disorders) | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Edema face (General disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fever (General disorders) | 1
Flushing (Vascular disorders) | 1
Gait disturbance (General disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Infusion related reaction (General disorders) | 1
Memory impairment (Nervous system disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Presyncope (Nervous system disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Tremor (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary frequency (Renal and urinary disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Sepsis (Infections and infestations) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Skin and subcutaneous disorder (Skin and subcutaneous tissue disorders) | 6
Endocrine Disorder (Endocrine disorders) | 1
Cardiac Disorder (Cardiac disorders) | 1
Infection and Infestation (Infections and infestations) | 1
Cold Sensitivity (Nervous system disorders) | 1
Surgical and Medical Procedure (Surgical and medical procedures) | 1
Cramping (Gastrointestinal disorders) | 1
Pseudo laryngospasm (Gastrointestinal disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT02918162/Prot_SAP_000.pdf